CLINICAL TRIAL: NCT07086430
Title: Independent Effects of Visceral Adipose Volume and Density on Patient Survival in Peritoneal Dialysis
Status: Completed | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Yue Qian, Principal investigator, RenJi Hospital
Other Study IDs: LY2025-017-B
Record Dates: First submitted 2025-07-14; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-04

CONDITIONS: Uremia; End Stage Renal Disease on Dialysis
Keywords: peritoneal dialysis; fat attenuation index on CT
MeSH Terms: conditions — Uremia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- derivation cohort; validation cohort

SUMMARY:
It was VAT volume predict patient outcome, while VAT density predicted baseline membrane function in PD patients and reflected peritoneal vascular density and local inflammation status.

ELIGIBILITY:
Inclusion Criteria:

* The study included peritoneal dialysis patients follow up in our center who had an abdominal CT scan within 2 weeks before PD catheter incubation.

Exclusion Criteria:

* Those with acute inflammation according to clinical signs, lab results or abdominal CT scan were excluded from the cohort.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study included peritoneal dialysis patients follow up in our center who had an abdominal CT scan within 2 weeks before PD catheter incubation. Those with acute inflammation according to clinical signs, lab results or abdominal CT scan were excluded from the cohort. In early years, abdominal CT scan was done if the patient reported history of abdominal abnormalities, such as history of cholelithiasis. Since 2020 it became a routine check before PD catheter incubation in our center. Those with cholelithiasis or hernia were suggested to had the preventive operation at the time of PD catheter incubation under general anesthesia. The patients started PD within 4 weeks after catheter incubation. A validation cohort was from a satellite center of the hospital. The inclusion criteria were same as the derivation cohort.
Sampling Method: Non-Probability Sample
Enrollment: 358 (Actual)
Dates: Start 2015-07-21 (Actual); Primary Completion 2023-07-11 (Actual); Study Completion 2025-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the association between peritoneal membrane solute transfer rate and abdominal visceral adipose tissue density measured on CT | from the baseline, 4 weeks before PD catheter insert surgery until patients quit PD or follow up up to 48 months